CLINICAL TRIAL: NCT04597437
Title: Zanamivir Treatment of Vascular Permeability in Dengue (ZAP-DENGUE): A Pilot Randomized Controlled Trial
Brief Title: Zanamivir Treatment of Vascular Permeability in Dengue (ZAP-DENGUE)
Acronym: ZAP-DENGUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Clinica de la Costa (Unknown); Global Disease Research (Unknown); Universidad Libre de Barranquilla (Unknown)
Responsible Party: Principal Investigator, Aileen Y Chang, PI, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCR203024
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue | interventions — Zanamivir

STUDY DESIGN:
Intervention Model Description: Pilot, randomized, double-blind, placebo-controlled trial of the safety and efficacy of inhaled zanamivir (n=37) versus placebo (n=37) therapy for dengue
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zanamivir (Experimental): In the treatment group, participants weighing less than 50 kg will receive 12 mg/kg and those weighing 50 kg and above will receive 600 mg as the initial dose intravenously every twelve hours for 5 days adjusted for renal function.
  Interventions: Drug: Zanamivir
- Placebo (Placebo Comparator): In the placebo group, participants will receive placebo normal saline solution intravenously every twelve hours for 5 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zanamivir — Intravenous zanamivir
  Arms: Zanamivir
Other: Placebo — In the placebo group, participants will receive placebo normal saline solution intravenously every twelve hours for 5 days.
  Arms: Placebo

SUMMARY:
ZAP-DENGUE is a pilot randomized, double-blind, placebo-controlled evaluation of the safety and efficacy of five days of intravenous zanamivir treatment to treat vascular permeability syndrome which is the main cause of death in dengue fever.

DETAILED DESCRIPTION:
ZAP-DENGUE is a pilot randomized, double-blind, placebo-controlled evaluation of the safety and efficacy of five days of intravenous zanamivir treatment to treat vascular permeability syndrome which is the main cause of death in dengue fever. Our central hypothesis is that zanamivir treatment is safe in patients with dengue infection, will significantly decrease serum sialic acid levels, and will result in fewer patients with the development of moderate or severe clinical plasma leakage. 74 male and non-pregnant female volunteers age 7 years and older from Colombia with a diagnosis of dengue fever with warning signs or severe dengue as per the World Health Organization 2009 definition with the presence of fever and positive rapid test for the presence of dengue non-structural protein-1 (NS1) will be randomized to zanamivir versus placebo. In the treatment group, all participants weighing less than 50 kg will receive 12 mg/kg and all participants weighing 50 kg and above will receive 600 mg as the initial dose intravenously every twelve hours for 5 days adjusted for renal function. In the placebo group, participants will receive placebo normal saline solution intravenously every twelve hours for 5 days.

All patients will receive blood draws for assessment of hematocrit, renal function, and biologic efficacy endpoints and clinical evaluation of signs and symptoms of vascular permeability (which may include ultrasound and radiograph) and adverse events daily during the five days of medication administration and once at follow up at 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged >7 years
4. Willingness to receive intravenous medication and be willing to adhere to the medication regimen
5. Have a diagnosis of dengue by dengue NS1 rapid test
6. Have had a self-informed fever >38 degrees C in the last 3 days.
7. Have dengue with warning signs as per the 2009 WHO criteria including one of the following: abdominal pain or tenderness, persistent vomiting, clinical fluid accumulation, mucosal bleeding, lethargy, restlessness, liver enlargement over 2 cm, augmented hematocrit, thrombocytopenia or severe dengue defined as dengue with severe plasma leakage leading to dengue shock and/or fluid accumulation with respiratory distress; severe hemorrhage; severe organ impairment (hepatic damage, renal impairment, cardiomyopathy, encephalopathy or encephalitis).
8. Enrollment in EPS (Entidadas Promotoras de Salud) or Sistema General de Seguridad Social en Salud (SGSSS)- Colombian Public Health Insurance.

Exclusion Criteria:

1. Pregnancy or lactation
2. Children in Care of the state
3. Patients who are unlikely to survive 48 hours
4. Unstable cardiac disease or arrhythmia at baseline
5. History of significant cardiac disease
6. Treatment with another investigational drug or other intervention within 1 month.
7. Encephalitis or unable to consent

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of intravenous zanamivir treatment versus placebo in dengue | Over 14 days
  Incidence of Treatment-Emergent Adverse Events will be assessed by daily active surveillance during drug administration and at 2-week follow-up as per the United States Food and Drug Administration guidelines.

SECONDARY OUTCOMES:
Levels of endothelial glycocalyx biomarkers in intravenous zanamivir treatment versus placebo in dengue | Over 14 days
  Serum concentration of key endothelial glycocalyx components due to endothelial damage such as sialic acid, heparan sulfate, and syndecan-1 will be assessed by ELISA.
  Serum concentration of sialidases (NEU2 and NEU3) that are directly inhibited by zanamivir will be assessed by ELISA.
Preliminary clinical efficacy of intravenous zanamivir treatment versus placebo in dengue | Over 14 days
  Presence of moderate or severe plasma leakage as defined by the Standard Clinical Endpoints for Use in Dengue Interventional Trials where moderate plasma leakage is defined as 15% change in hematocrit or evidence of fluid on ultrasound or X-ray and severe plasma leakage is defined at the presence of shock or respiratory compromise with evidence of plasma leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Chang, MD, Principal Investigator — George Washington University
Locations (2):
- Colombia (2):
  - Cien Salud IPS SAS, Barranquilla, Atlántico
  - Clinica de la Costa SAS, Barranquilla, Colombia

IPD SHARING:
Plan to Share IPD: No
De-identified information can be shared with other investigators. Please contact Dr. Aileen Chang at chang@email.gwu.edu